CLINICAL TRIAL: NCT04601961
Title: Effects of Mode of Anaesthesia on Circulating Tumour Cells in Patients Undergoing Inhalational Versus Total Intravenous Anaesthesia for Hepatocellular Carcinoma Surgery : A Randomised Controlled Trial
Brief Title: Effects of TIVA Versus Inhalational Anaesthesia on Circulating Tumour Cells in Hepatocellular Carcinoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UW 20-022
Record Dates: First submitted 2020-09-21; First posted 2020-10-26 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Circulating Tumor Cell; Hepatocellular Carcinoma
Keywords: Circulating Tumor Cell; Hepatocellular Carcinoma; anaesthesia; TIVA; SEVO
MeSH Terms: conditions — Neoplastic Cells, Circulating; Carcinoma, Hepatocellular | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEVO Group (Active Comparator): Patients in SEVO group will be anaesthetized by inhalational anaesthesia using sevoflurane.
  Interventions: Drug: Sevoflurane
- TIVA group (Experimental): The patients in TIVA group will be anaesthetized using total intravenous propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Monitoring and other anaesthetic procedures including the management of hypertension and hypotension will be the same as SEVO group. Induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Sevoflurane will not be used, and oxygen and air would be given to provide a FiO2 of 30-50%.
  Target controlled infusion (TCI) with a modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia and titrated to effect. The usual effect site concentration is 1.5-3 mcg.ml-1 and BIS monitoring will also be used to produce a value of between 40-60. As with patients in the SEVO group, remifentanil will be infused at a rate of between 0.1-0.3 mcg.kg.min-1.
  Arms: TIVA group
Drug: Sevoflurane — Propofol 1.5-3mg/kg, remifentanil 1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be used intravenously for induction of general anaesthesia. Intubation would be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane, air and oxygen will be used for maintenance of general anaesthesia. FiO2 will be kept between 35-50%. BIS monitoring will be applied and level of anaesthetia will be titrated to maintain a BIS value of between 40-60. Intravenous remifentanil infusion between 0.1-0.2 mcg/kg/min will be given and this will be titrated to provide optimal haemodynamic parameters.
  Arms: SEVO Group

SUMMARY:
More than 80% of patients with cancer will be exposed to anaesthesia at some point in their treatment. There is increasing evidence that perioperative events, including the type of anaesthesia drugs utilised, have an impact on cancer recurrence and metastases.

Although potentially and theoretically curative, surgical resection, manipulation and trauma may disseminate tumour cells and reduce immunity. There have been a number of suggestions as to why cancer may be, paradoxically, worsened by surgery and what methods may be used to mitigate this. One of these is propofol based total intravenous anaesthesia (TIVA), whereby the traditional inhalational anaesthetic drugs are avoided. Commonly used inhalational drugs, such as sevoflurane and desflurane, are pro-inflammatory.

Propofol, however, has anti-inflammatory and anti-oxidative properties, induces apoptosis and has specific inhibitory effects on tumour cell growth in vitro. Laboratory investigations, animal models, retrospective clinical studies and initial clinical research are producing evidence that inhalational anaesthesia facilitates tumour recurrence and metastasis, whilst TIVA can prolong survival.

This randomised, controlled trial will look at the effects on DNA damage and biomarkers of immunity and inflammation of inhalational anaesthesia versus TIVA in patients undergoing surgery for hepatocellular carcinoma, a common tumour in the Southern Chinese population, for whom surgery is potentially-curative. It will focus on subjects undergoing open and laparoscopic hepatectomy and investigate changes in biomarkers of inflammation, immunity and gene expression from the patients' blood samples taken before, during and after surgery.

Patients will also be followed-up for cancer recurrence, morbidity and five-year mortality. Results could represent a breakthrough in knowledge of how anaesthetic agents impact the results of cancer surgery, and have important implications for a more disease- sensitive approach to improving management and outcomes in these patients.

DETAILED DESCRIPTION:
Pre-operative care

Pre-operative assessment will be performed at the preadmission clinic or at the general ward. Patients will be fasted for intake of solid food for 6 hours and clear liquids for 2 hours. Sedative premedication will not be prescribed.

Anaesthesia and intraoperative care

SEVO Group

Patients from the SEVO group will be anaesthetized according to the following protocol:

On arrival at the operation theatre, an intravenous cannula will be inserted. Standard monitoring with pulse oximeter, non-invasive blood pressure, and three-lead electrocardiogram will be applied prior to induction. Non-invasive blood pressure (NIBP) will be checked at least every 5 minutes throughout the operation. An arterial line may be inserted at the discretion of the anaesthetist before or after induction, with invasive blood pressure monitoring in lieu of NIBP if deemed necessary. Additional intravenous cannulas or central lines may also be inserted to facilitate fluid therapy, measure the central venous pressure or administer drugs, also at the discretion of the attending anaesthetist.

Anaesthesia will be induced with titrated, manual propofol injection of 1-2 mg.kg-1. Remifentanil infusion will be given for analgesia at a rate of 0.1 - 0.35 mcg.kg.min-1 as required, according to haemodynamic parameters. Cisatracurium 0.15 mg.kg-1 or atracurium 0.5 mg.kg-1 will be used for muscle relaxation. Tracheal Intubation will be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane at 0.5- 1 MAC, air and oxygen will be used for maintenance of general anaesthesia. Processed EEG (BIS™) will be utilized to monitor depth of anaesthesia, aiming at a BIS value of 40-60. FiO2 will be kept between 35-50% to maintain and SaO2 of > 95%. Further muscle relaxants can be given during the operation if required.

In accordance with British consensus guidelines on intravenous fluid therapy for Adult Surgical Patients [22], intraoperative fluid or blood loss will be initially replaced with balanced crystalloid solution, preferably Plasmalyte A (a physiologically balanced electrolyte solution similar to extracellular fluid), for up to 20% of body volume, with additional fluid replacement with colloid or crystalloid at the discretion of the anaesthetist. Intravenous phenylephrine, ephedrine or fluid administration may also be given for management of hypotension. Intravenous anti-hypertensive agents such as beta blockers (e.g. esmolol, labetalol) and glyceryl trinitrate can be given if hypertension occurs.

Patients will receive standardized opioid analgesia of 0.1 mg.kg-1 intravenous morphine intra-operatively followed by patient-controlled analgesia (PCA) morphine post-operatively, as well as local anaesthesia (0.5% levobupivacaine) injected in the areas of surgical incision during wound closure for pain control.

Forced air warming blankets will be used with the aim of keeping a core temperature of 35.5-37.5 degrees Celsius. Ondansetron 4mg IV will be given 30 minutes before end of surgery.

Sevoflurane and remifentanil infusion will be switched off at the end of the procedure. Reversal of muscle relaxation can be achieved if required with neostigmine 50 mcg.kg-1 IV and atropine 20 mcg.kg-1 IV. Patients will subsequently be transferred to the post anaesthetic care unit (PACU) for monitoring for at least 30 minutes.

TIVA Group

Patients in the TIVA group will be anaesthetized according to the following protocol:

Monitoring and other anaesthetic procedures including the management of hypertension and hypotension will be the same as SEVO group. Induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Sevoflurane will not be used, and oxygen and air would be given to provide a FiO2 of 30-50%.

Target controlled infusion (TCI) with a modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia and titrated to effect. The usual effect site concentration is 1.5-3 mcg.ml-1 and BIS monitoring will also be used to produce a value of between 40-60. As with patients in the SEVO group, remifentanil will be infused at a rate of between 0.1-0.3 mcg.kg.min-1.

Post-operative care for both groups In the recovery room after surgery, numerical rating pain score (NRS) will be used to assess level of pain. Patients will select a whole number (0-10 integers) that best reflects the intensity of his/her pain, in which 10 represents the maximal imaginable pain. Boluses of 2 mg intravenous morphine will be given every 5 minutes until the numerical rating scale (NRS) is less than or equal to 4/10. A patient controlled analgesia (PCA) machine will then be connected. The machine will be configured to give 1 mg of morphine whenever the patient demands with the lockout duration set to 5 minutes. No background infusion will be given and the maximum dose limit will be 0.1 mg.kg-1 per hour of morphine.

On post-operative day 1, when the patient resumes a fluid diet, oral celecoxib 200 mg will be given twice daily for 3 days.

Whilst on PCA morphine, the patient's respiratory rate, oxygen saturation (SpO2) and sedation score will be monitored every hour. Heart rate and blood pressure will be checked every 4 hours. NRS pain scores at rest and during cough/movement, cumulative PCA morphine doses, and number of PCA demands/goods delivered, and side effects (nausea, vomiting, dizziness, hypotension, desaturation) will be recorded every 4 hours. Patients will be assessed by a "pain team" every day to determine sufficiency of analgesia, as per usual practice.

Patients will be kept on PCA morphine for at least 2 days. If NRS pain scores during cough/ movement on postoperative day 2 are less than or equal to 3/10, PCA morphine will be stopped. PCA morphine will be continued if NRS is equal or greater than 4, or if the patient remains on a high PCA use. Assessment for analgesia will be conducted daily. Evaluation for complications will be required if NRS pain score is 4 or higher on postoperative day 5. The patient will be further managed at the discretion of the anaesthetist.

After PCA morphine has been withdrawn, NRS pain scores at rest and during cough/ movement, as well as the dose and frequency of rescue analgesia used will be charted once a day until discharge.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18-80 years old with primary hepatocellular carcinoma presenting for elective open hepatectomy surgery in Queen Mary Hospital, Hong Kong, will be invited to join this randomised, controlled trial.

Exclusion Criteria:

Pre-operative factors

* Contraindication to general anaesthesia
* Autoimmune / Chronic inflammatory diseases e.g. Systemic Lupus Erythematosus (SLE), Rheumatoid Arthritis(RA) etc.
* Chemotherapy in the past year
* Steroid therapy
* Surgery for tumour removal in the past year
* patients post liver transplantation Intra-operative factors
* Regional Anaesthesia

Administration of:

* Nitrous oxide
* Inhalational agents (with the exception of sevoflurane)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
HIF-1 gene expression | 24 hour
  the detection of a two-fold difference between the pre-operative blood sample and 24-hour post-operative blood sample in HIF-1 gene expression in the SEVO group, and a less than two-fold difference in the same samples of the TIVA group

SECONDARY OUTCOMES:
Change in number of recurrence | 2 year
  Change in the incidence of two-year recurrence between TIVA and SEVO group
Level of Gene expression | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of Gene expression (HIF-1, IL-6, TNF-alpha) will be measured from the RNA/cDNA extracted from blood sample taken at different timepoints by Polymerase chain reaction test
Level of DNA damage | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of DNA damage will be measured from the white blood cells extracted from blood sample taken at different timepoints by Comet Assay test
Level of C-reactive protein | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of C-reactive protein will be measured from the Plasma extracted from blood sample taken at different timepoints by Commercial Kit
Level of Glutathione Peroxidase | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of Glutathione Peroxidase will be measured from the Red blood cells extracted from blood sample taken at different timepoints by Commercial Kit
Level of Superoxide dismutase | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of Superoxide dismutase will be measured from the Red blood cells extracted from blood sample taken at different timepoints by Commercial Kit
Level of Oxidative damage DNA | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of Oxidative damage DNA (8-oxoGuo, 8-oxodG) will be measured from the Plasma extracted by Commercial Kit
Level of tumor necrosis factor | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The level of tumor necrosis factor (IL-6, TNF-alpha, HIF-1) will be measured from the Plasma extracted by An enzyme-linked immunosorbent assay (ELISA)
Number of Circulating tumour cells | Pre-operative, Intra-operative, Immediately post-operative and 24 hours post-surgery
  The number of Circulating tumour cells will be isolated from the blood samples taken at different timepoints by filtration and count under microscope

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Irwin, M.B. Ch.B, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Li Ka Shing Faculty of Medicine, Hong Kong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04601961/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04601961/ICF_001.pdf